CLINICAL TRIAL: NCT00786396
Title: Directly Observed Therapy for Community-Released HIV+ Prisoners
Acronym: Connect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01 DA 0179059
Record Dates: First submitted 2008-11-05; First posted 2008-11-06 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: HIV/AIDS; Substance Abuse
Keywords: HIV; AIDS; substance abuse; directly administered antiretroviral therapy; adherence; Substance Abuse and Dependency
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DAART (Experimental): Group that will be observed daily taking their medications for a period of six months. Followed by the remaining six months of the intervention in which the subject will take medications on their own.
  Interventions: Behavioral: Directly administered antiretroviral therapy
- 2 (No Intervention): SAT (standard of care) group will take their medications as directed by their physicians for the period of one year.

INTERVENTIONS:
Behavioral: Directly administered antiretroviral therapy — Daily observation of subjects taking their HIV medications
  Arms: DAART

SUMMARY:
The aim of this study is to develop effective interventions for HIV-infected prisoners who are released to the community. The intervention that we will study will be directly observed therapy (DAART/DOT) and we will compare this to the current standard of care that involves self-administered therapy (SAT). All subjects will get transitional case management and all subjects with a prior history of opiate dependence will be offered opiate substitution therapy (buprenorphine or methadone).

Hypotheses:

* At the end of six months those receiving DAART will have a higher level of adherence to HAART as compared to the SAT group.
* The DAART Intervention will result in subjects having lower viral loads and higher CD4 counts as compared to the SAT group.
* At the end of six months, the DAART group will have a lower rate of recidivism to jail/prison as compared to the SAT group.
* Over the year, the DAART group will be more likely to make repeated primary HIV care visits than the SAT group.

DETAILED DESCRIPTION:
Any individual that is HIV positive and incarcerated for at least a period of 90 days and on antiretroviral medications would be referred to the study by the medical staff of the incarceration facilities prior to release or within 30 days of release an individual would be able to self refer.

Subjects would be screened and consented and interviewed prior to their release from incarceration, on their day of release, and monthly for a period of one year. At the time of their day of release interview, subjects are randomized to either the intervention DAART group or the standard of care SAT group. All subjects would be assessed and offered opiate substitution therapy if there was a prior history of opiate dependency as a means of relapse prevention.

Subjects in DAART would be seen everyday for a period of six months by a team of research assistants who observe the subjects taking their medications, and their last six months would be done as standard of care. Standard of care SAT subjects would continue to take their medications on their own as prescribed. All subjects would be interviewed monthly and quarterly would have laboratory blood tests completed.

ELIGIBILITY:
Inclusion Criteria:

* HIV seropositive
* 18 years of age or older
* incarcerated for a minimum of 90days
* living in New Haven or Hartford
* currently on HAART or willing to begin HAART medications

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2004-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Virological success, defined as greater than 1 log HIV-1 copies/mL reduction or Viral load less than 400 copies/mL at the end of six months on the intervention. | 12 months

SECONDARY OUTCOMES:
DAART subjects will be more likely to make primary HIV care visits than those receiving SAT. | 12
Lower rate of recidivism and to illicit drug use | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederick L Altice, MD, Principal Investigator — Yale University; Gerald Friedland, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Yale University-Yale Clinical Research, Hartford, Connecticut
  - Yale University School of Medicine, New Haven, Connecticut

REFERENCES:
- [Background] Saber-Tehrani AS, Springer SA, Qiu J, Herme M, Wickersham J, Altice FL. Rationale, study design and sample characteristics of a randomized controlled trial of directly administered antiretroviral therapy for HIV-infected prisoners transitioning to the community - a potential conduit to improved HIV treatment outcomes. Contemp Clin Trials. 2012 Mar;33(2):436-44. doi: 10.1016/j.cct.2011.11.002. Epub 2011 Nov 12. PMID 22101218
- [Background] Springer SA, Chen S, Altice F. Depression and symptomatic response among HIV-infected drug users enrolled in a randomized controlled trial of directly administered antiretroviral therapy. AIDS Care. 2009 Aug;21(8):976-83. doi: 10.1080/09540120802657555. PMID 20024753
- [Background] Springer SA, Chen S, Altice FL. Improved HIV and substance abuse treatment outcomes for released HIV-infected prisoners: the impact of buprenorphine treatment. J Urban Health. 2010 Jul;87(4):592-602. doi: 10.1007/s11524-010-9438-4. PMID 20177974
- [Background] Meyer JP, Qiu J, Chen NE, Larkin GL, Altice FL. Emergency department use by released prisoners with HIV: an observational longitudinal study. PLoS One. 2012;7(8):e42416. doi: 10.1371/journal.pone.0042416. Epub 2012 Aug 3. PMID 22879972